CLINICAL TRIAL: NCT03594292
Title: Clinical Study of MedShape FASTFORWARDTM Bunion Correction System in Treating Hallux Valgus Patients
Brief Title: FASTFORWARDTM Bunion Correction System in Treating Hallux Valgus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung Kuo, Attending Physician, Department of Orthopedics, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH105-REC2-075
Record Dates: First submitted 2018-06-24; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-01

CONDITIONS: Hallux Valgus and Bunion (Disorder)
Keywords: hallux valgus and Bunion
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FASTFORWARDTM Bunion (Experimental): The participants are treated with FASTFORWARDTM Bunion Correction system. The FASTFORWARDTM Bunion Correction system employed 3D printed titanium bone tether plate at second metatarsal. Due to the merit of 3D printing technology, the plate is designed to broadly distribute forces across bone to secure mechanical integrity of the bone. The FASTFORWARDTM Bunion Correction system has been cleared by the United States Food and Drug Administration.
  Interventions: Device: FASTFORWARDTM Bunion
- Conventional Surgery (Active Comparator): The participants are treated with fusion surgery. This procedures is a standard treatment for 1st metatarsal hallux valgus by cutting, realigning and fusing the 1st metatarsal or fusing the metatarsal-cuneiform joint.
  Interventions: Procedure: Conventional surgery

INTERVENTIONS:
Device: FASTFORWARDTM Bunion — The participants will be assign to implantation of FASTFORWARDTM Bunion correction system surgery as a experimental group.
  Arms: FASTFORWARDTM Bunion
Procedure: Conventional surgery — The participants will assign to conventional surgery as a control group, the procedure is a standard treatment for the 1st metatarsal hallux valgus.
  Arms: Conventional Surgery

SUMMARY:
The FASTFORWARDTM Bunion Correction system has been cleared by the United States Food and Drug Administration for sale. This study is to investigate the clinical outcome of MedShape FASTFORWARDTM Bunion Correction system in treating hallux valgus patients at CMUH.

Criteria-There will be 12 subjects with a painful bunion and hallux valgus between 20 and 65 years of age and an adequate range of movement. Patients with rheumatoid arthritis, failed previous hallux valgus surgery and symptomatic and/or radiological arthritis of the MTP joint will be excluded.

Protocol-The PI and SC explain the detail and purpose of the project to the patient to the language to the patient is comfortable with. The explanation has to be at least 1 hour. Be sure the patients understand the full detail before the surgery.

Computer tomography scan, gait analysis and blood biochemical analysis will be taken in 1-2 weeks after patient is enrolled in the subject. Before surgery, the titration bone tether plate designed to match patent's second metatarsal contour will be manufactured using 3D printing technology. Printed titanium plate and PEEK screws used to secure tethering suture tape in the first metatarsal will be sterilized prior implantation. The surgery time, recovery period and effectiveness after implantation will be recorded. To observing the recovery situation, patients will back to out-patient clinic at 1st, 2nd, 3rd, 4th, 6th, 12th, 24th weeks. During these period, physical examination, wound dressing, VAS, X-ray scan will be arranged. The detail arrangements below:

1.1st week: physical examination, wound dressing, VAS

2.2nd week: physical examination, wound dressing, VAS

3.3rd week: physical examination, wound dressing, VAS, X-ray scan, remove stiches

4.4th week: physical examination, VAS

5.6th week: physical examination, VAS, X-ray scan

6.12th week: physical examination, VAS, X-ray scan

7.24th week: physical examination, VAS, X-ray scan, CT scan, gait analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with a painful bunion and hallux valgus between 20 and 65 years of age and an adequate range of movement

Exclusion Criteria:

* Patients with rheumatoid arthritis, failed previous hallux valgus surgery and symptomatic and/or radio-logical arthritis of the MTP joint

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Intermetatarsal 1-2 angle postoperative | 6 month
  Evaluating the angle among the 1st and the 2nd metatarsal assess by X-ray scan and CT scan

SECONDARY OUTCOMES:
Assessment Foot Pressure | 6 month
  Foot pressure assess by gait analysis
Pain using a visual analog scale | 6 month
  Evaluating pain level by using visual analog scale
Intermetatarsal 1-2 angle | 6 month
  Evaluating the angle among the first metatarsal and the first phalanx assess by X-ray scan

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Kuo, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Beitun District, Taiwan

IPD SHARING:
Plan to Share IPD: No